CLINICAL TRIAL: NCT06760117
Title: Phase I Study of Irinotecan Dose Adjustment Guided by UGT1A1*6 Genotype in VIT Regimen for the Treatment of Relapsed and Refractory Childhood Solid Tumors
Brief Title: UGT1A1 Genotype-drien Phase I Study of Irinotecan in VIT Regimen for the Treatment of Pediatric R/R Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Prof, Sun Yat-sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Sun Yat-sen University Cancer
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Solid Tumor
Keywords: UGT1A1 gene; irinotecan
MeSH Terms: interventions — Irinotecan; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia (Experimental): A phase Ia dose escalation study of temozolomide and vincristine at fixed doses and escalating doses of irinotecan (patients with wild-type UGT1A1 *6 (T/T) genotype are eligible for dose escalation of irinotecan) for the treatment of relapsed/refractory pediatric solid tumors. The standard 3+3 patient enrollment design was adopted.
  Interventions: Drug: Irinotecan (CPT-11); Drug: Temozolomide (TMZ); Drug: Vincristine
- Phase Ib (Other): In the VIT regimen, irinotecan will be administered using the RP2D dose determined by Phase Ia, with an expansion to 9-12 additional patients to further explore efficacy and safety.
  Interventions: Drug: Irinotecan (CPT-11); Drug: Temozolomide (TMZ); Drug: Vincristine

INTERVENTIONS:
Drug: Irinotecan (CPT-11) — Irinotecan will start at a dose of 50mg/m² and escalate to explore the maximum tolerated dose.
Drug: Temozolomide (TMZ) — TMZ：100mg/m2/d，d1-5
Drug: Vincristine — VCR: 1.5mg/m2/d(≯2mg), d1

SUMMARY:
Irinotecan is a commonly used salvage chemotherapy drug for children with relapsed and refractory solid tumors. Common dose-limiting toxicities of irinotecan include abdominal pain and diarrhea. Studies have shown that patients with UGT1A16 gene mutations have a higher incidence of these side effects, thereby limiting the dosage of irinotecan. The combination of irinotecan with temozolomide and vincristine is a common salvage chemotherapy regimen for children with relapsed and refractory solid tumors. Currently, the recommended dose of irinotecan is 50mg/m², but there is still significant room for improvement in the efficacy of VIT for these children. Whether patients with wild-type UGT1A16 can further increase the dosage of irinotecan, thereby enhancing the efficacy of the VIT regimen, is the focus of our research.

DETAILED DESCRIPTION:
Children with relapsed and refractory solid tumors and wild-type UGT1A1 gene are enrolled in this study. The doses of temozolomide and vincristine are fixed, while irinotecan in the VIT regimen begins at a starting dose of 50mg/m² and escalates across five dosage groups, with the highest dose group being 110mg/m². This study aims to determine the maximum tolerated dose of irinotecan and the safety of incremental irinotecan dosing, as well as the objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS). This will lay the foundation for future Phase II/III clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years.
2. Relapsed and refractory childhood solid tumors (pathologically confirmed). Definition of relapsed and refractory patients: 1. Patients who fail to achieve GPR or CR after first-line treatment are defined as refractory; 2. Patients who achieve CR after first-line treatment but relapse after more than 1 month are defined as relapsed.
3. Must have undergone UGT1A1*6 genotype testing (provided free of charge by Jiangsu Hengrui Medicine Co., Ltd.), with results being wild type (T/T).
4. Patients must be at least 3 weeks post the last myelosuppressive chemotherapy and at least 6 months post hematopoietic stem cell transplantation, 2 weeks post local radiotherapy, 6 months post craniospinal or extensive pelvic radiotherapy, or 6 weeks post extensive bone marrow radiotherapy.
5. Must have at least one measurable lesion as defined by RECIST criteria;
6. Karnofsky score (for ages > 10, see Annex I) or Lansky score (for ages ≤ 10, see Annex II) ≥ 50 points;
7. Expected survival time ≥ 6 months;
8. Patients must have fully recovered from all acute toxic effects of previous anticancer chemotherapy: a) Bone marrow suppression chemotherapy: at least 21 days post the last bone marrow suppressive chemotherapy; b) Hematopoietic growth factors: at least 14 days post the last dose of long-acting growth factor or 7 days post the last dose of short-acting growth factor;
9. For patients known not to involve the BM: a) Absolute neutrophil count (ANC) ≥ 1.0×10⁹/L; b) Non-transfused platelet count ≥ 100.0×10⁹/L; c) Hemoglobin ≥ 80 g/L;
10. Liver and kidney functions must meet the following criteria: a) Total bilirubin (conjugated + unconjugated) ≤ 1.5× upper limit of normal (ULN) for age; b) Aspartate aminotransferase (AST) ≤ 2.5×ULN (≤ 110 U/L); c) Glomerular filtration rate or creatinine clearance ≥ 70 mL/min/1.73 m² or corresponding age-normal serum creatinine; d) Serum albumin ≥ 20 g/L.
11. Capable of adhering to outpatient treatment, laboratory monitoring, and necessary clinical visits during the study period;
12. Parents/guardians of children or adolescent subjects must be able to understand, consent to, and sign the informed consent form (ICF) and applicable child consent forms before initiating any protocol-related procedures; if parents/guardians agree, subjects must be capable of expressing consent (when applicable).

Exclusion Criteria:

1. Patients who have previously received chemotherapy with irinotecan combined with temozolomide and vincristine, or patients who have progressed after receiving treatment with irinotecan or temozolomide;
2. Patients receiving P450 enzyme-inducing antiepileptic drugs (antiepileptic drugs affect the clearance of irinotecan);
3. During the study period, patients must not receive any other chemotherapy, radiotherapy, or granulocyte colony-stimulating therapy;
4. Patients positive for hepatitis B surface antigen;
5. Patients infected with HIV or syphilis;
6. Patients who have previously undergone organ transplantation;
7. Uncontrolled active systemic bacterial, viral, or fungal infections; Clostridium difficile infection requiring treatment;
8. Patients allergic to dacarbazine or cephalosporin drugs;
9. Patients requiring high-dose dexamethasone treatment;
10. Patients with a severe history of neurological or psychiatric disorders, including epilepsy or autism.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MTD and DLT | From the start of the VIT regimen to 16 days after the end of the regimen.
  The maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of irinotecan

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — SunYat Sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No